CLINICAL TRIAL: NCT00847977
Title: Intérêt d'Utiliser Des solutés de Remplissage équilibrés à la Phase précoce d'un Traumatisme crânien Grave Pour Limiter l'Acidose hyperchlorémique
Brief Title: Interest of Using Balanced Fluid for Infusion at the Early Phase of an Acute Cranial Trauma for Limiting Hyperchloremic Acidosis
Acronym: IsoTC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Cellule de Promotion de la Recherche Clinique, CHU de Nantes
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BRD 08/3-J
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Head Trauma
Keywords: Acute head trauma
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Heafusine - Physiologic serum
  Interventions: Drug: use of a non balced fluid and of a macromolecular fluid
- 2 (Experimental): Isofundine - Tetraspan
  Interventions: Drug: use of balanced crystalloids fluid and macromolecular fluid

INTERVENTIONS:
Drug: use of a non balced fluid and of a macromolecular fluid — Physiological serum: basic flow 30 ml/kg/j during 48 hoursand boli wished by physicians 20 ml/kg on 20 minutes Heafusine: boli 10 ml/kg on 20 minutes
  Other Names: Physiological serum and HEAfusine
  Arms: 1
Drug: use of balanced crystalloids fluid and macromolecular fluid — Isofundine: basic flow 30 ml/kg/j during 48 hoursand boli wished by physicians 20 ml/kg on 20 minutes Tetraspan: boli 10 ml/kg on 20 minutes
  Other Names: Tetraspan - Isofundine
  Arms: 2

SUMMARY:
isotonic NaCl serum is the first intent solution for infusion during the initial phase of reanimation for an acute cranial traumatism.

However, its use can trigger an hyperchloremic metabolic acidosis, what could be deleterious for the future of this patient.

Isofundine present all charateristics to be use in this indication: pharmacokinetic and pharmacodynamic similar to the physiologic serum, iso-osmolarity to plasma, no glucose provision and no interaction with hemostasis.

DETAILED DESCRIPTION:
Participation in the study lasts 7 days per patient.

Both solutions are crystalloids who received MA in France for ISOFUNDINE, MA in Germany with pending MA in France for TETRASPAN, including an indication for infusion. Both solutions are consistent with the recommendations of intensive care of a traumatized brain: iso-osmolar and without glucose. The study is an emergency: the resuscitation of a head injury, for which the plasma by crystalloids may be delayed.

J0: Day of Inclusion

On arrival at the emergency operating room at the diagnosis of a serious head injury alone, the anaesthetist that supports the patient in an initial phase includes the patient in the study.

A H0, it is holding the patient randomization and continued his rehabilitation with the lot of fluids allocated. If he wants to use macro-molecules, it may use HydroxyEhtylAmidons(HEA). Each batch assigned to a patient includes a crystalloids and HEA: witnesses arm includes saline solution and the HEAfusine while the interventional arm includes Isofundine and tetraspan. These treatment are indistinguishable and both provided by the laboratory Braun. They will be kept in operating emergency to be the most readily available, upon arrival of the patient. If the health of the patient requires a refill crystalloids emergency even before randomization did not take place, the clinician uses originally Saline and starts the protocol as soon as possible as soon as the patient him can take the few minutes needed to achieve inclusion. The first biological assessment include the determination of natremia, of kaliemia, of magnesemia, the ionized calcium, the lactatemia of albumin, the osmolarity of plasma and blood gases. These strengths are in Biological standard of care of a traumatized brain.

Apart from the contribution of crystalloids, the rest is therapeutic to the discretion of clinicians. The indication of monitoring the intra-cranial pressure sensor intra-parenchymatous is left to the discretion of the clinician without obligation associated with the study. As requires the usual care of this pathology, the patient is then transferred to intensive care.

J1 and J2

In accordance with the Memorandum of service, a basic daily infusion of crystalloids (30 ml / kg / day) is prescribed to all patients during the first 48 hours. The crystalloids used for these basic inputs is the lot assigned at inclusion.

If the indications of plasma referred to by hemodynamic boli solutes remain free indication of the doctor taking care of the patient, type of fluid used is the batch assigned to the patient (Isofundine-Physiologic serum), including the use of macromolecules that are available in the lot assigned to the patient (Heafusine-tetraspan).

Biological monitoring TBI usually based on a biological assessment every 12 hours. It includes a ionograms blood and blood gases. On the same samples without extract a larger volume of blood, we collect specifically in biological assessments:

* ionized calcium, magnesemia, natremia, kaliemia.
* lactatemia.
* albumin.
* plasma osmolarity. No blood gases.

Neurological based monitoring as requested by the clinician is changing the values of either the PIC transcranial doppler.

The contribution of treatment under study stops at the 48th hour, after that time, the inflow of fluid is pursued in accordance with the wishes of doctors, and the type of product is imposed by the study .

J7 or exit resuscitation

The end of the study is the 7th day of inclusion (not trauma), or the day of release resuscitation if it precedes the 7th day. This is the end of the collection of clinical data and biological weapons. From J2-J7, no treatment and no record is imposed by the study. This is a simple monitoring period assessing the future clinical neurological patients.

ELIGIBILITY:
Inclusion Criteria:

* Glasgow < or equal to 8
* Patient > 18 years old

Exclusion Criteria:

* Polytraumatism
* Pregnancy
* Patient under guardianship
* renal insufficiency, hypokaliemia, hypocalcemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Incidence of hyperchloremic acidosis during the 2 first days of acute cranial traumatism. | J1 and J2

SECONDARY OUTCOMES:
Incidence of hypokaliemia and hypocalcemia | J1 and J2
Study of treatment effect on the evolution of intracranil pressure. | J1 and J2

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Réanimation CHU de Nantes Boulevard Jean Monnet, Nantes, France

REFERENCES:
- [Derived] Roquilly A, Loutrel O, Cinotti R, Rosenczweig E, Flet L, Mahe PJ, Dumont R, Marie Chupin A, Peneau C, Lejus C, Blanloeil Y, Volteau C, Asehnoune K. Balanced versus chloride-rich solutions for fluid resuscitation in brain-injured patients: a randomised double-blind pilot study. Crit Care. 2013 Apr 19;17(2):R77. doi: 10.1186/cc12686. PMID 23601796